CLINICAL TRIAL: NCT00413426
Title: An Open-labeled, Randomized, Single Dose, Three Period, 2-sequence Crossover Study to Investigate the Pharmacokinetics of Darifenacin When Given as 7.5 mg Oral Doses of a Modified Release Suspension, as Compared to the Commercial Modified Release Tablet in Healthy Adult
Brief Title: Study to Compare How the Body Changes the Blood Level of Darifenacin Tablet Form vs. the Modified Release Liquid Form in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Procter and Gamble (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CDAR328B2101
Record Dates: First submitted 2006-12-18; First posted 2006-12-19 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Pharmacokinetics; oral; single dose; table; suspension; release; darifenacin; healthy subjects; Healthy volunteers study
MeSH Terms: interventions — darifenacin

INTERVENTIONS:
Drug: Darifenacin (DAR328)

SUMMARY:
This purpose of this study is to compare the how the body changes the blood level of a single dose of darifenacin when given as 7.5 mg modified release tablet and the modified release liquid suspension (1.5 mg/ml) under fasted and fed conditions in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, male or female subjects age 18 to 50 years of age (inclusive)
* In good health
* Female subjects either surgically sterilized at least 6 months prior to study participation or post-menopausal (no regular menstrual bleeding for at least 2 years)
* Body mass index within the range of 18.5 to 29.9 kg/m2 and weigh at least 45 kg

Exclusion Criteria:

* Smokers
* History of
* Urinary retention, narrow-angle glaucoma, myasthenia gravis, severe hepatic impairment, severe ulcerative colitis, toxic megacolon
* Symptomatic hiatus hernia, erosive or symptomatic gastroesophageal reflux disease/heartburn (>2 days in a week), severe constipation, gastrointestinal obstructive disorders, and gastric retention.
* Clinically significant cardiac abnormalities, fainting, low blood pressure upon standing, irregular heartbeats
* Acute or chronic bronchospastic disease (including asthma and chronic obstructive pulmonary disease)
* Clinically significant drug allergy or history of atopic allergy (asthma, urticaria, eczematous dermatitis)
* Known hypersensitivity or severe adverse event to darifenacin or similar drugs
* Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs or which may jeopardize participation in the study
* Immunodeficiency diseases, including a positive HIV (ELISA and Western blot) test result
* Positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result.
* Drug or alcohol abuse within the 6 months prior to dosing
* Use of prescription drugs within 4 weeks prior dosing, or over-the-counter medication (vitamins, herbal supplements, dietary supplements) within 2 weeks prior to dosing. Paracetamol is acceptable.
* Participation in any clinical investigation within 4 weeks prior to dosing
* Donation or loss of 400 mL or more of blood within 8 weeks prior to dosing.
* Significant illness within 2 weeks prior to dosing.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28
Dates: Start 2006-06; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Comparison of the PK of a single dose of 7.5 reference modified release tablet of darifenacin and the tested modified release liquid suspension (1.5 mg/ml) of darifenacin under fasted conditions in healthy subjects
Comparison of the PK of a single dose of darifenacin when given as an oral dose of a 7.5 mg modified release liquid suspension in the fed and fasted states

SECONDARY OUTCOMES:
Safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Principal Investigator — Investigator site
Locations (1):
- Novartis Investigative Site, Mumbai, India